CLINICAL TRIAL: NCT02626650
Title: Recent Experiences and Presentation Format: Study of Concussion Symptom Elicitation
Brief Title: Recent Experiences With Concussions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Carnegie Mellon University (Other); University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: HS15-334
Record Dates: First submitted 2015-12-04; First posted 2015-12-10 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Check symptoms one has experienced (Active Comparator): This is the baseline condition. When asked to indicate concussion symptoms (or most other kinds of symptoms for medical conditions), people usually place a check mark next to each symptom they have experienced.
  Interventions: Other: Symptom elicitiation
- Check symptoms one has not experienced (Experimental): Participants place a check mark next to each symptom they have NOT experienced in the most recent sports season.
  Interventions: Other: Symptom elicitiation
- Uncheck symptoms one has experienced (Experimental): To begin, all symptoms will be automatically checked. Participants are told to remove a check mark from each symptom they have experienced in the most recent sports season.
  Interventions: Other: Symptom elicitiation
- Uncheck symptoms one has not experienced. (Experimental): To begin, all symptoms will be automatically checked. Participants are told to remove a check mark from each symptom they have NOT experienced in the most recent sports season.
  Interventions: Other: Symptom elicitiation

INTERVENTIONS:
Other: Symptom elicitiation — Survey procedure, people check or uncheck symptoms they have or haven't experienced. We randomly assign participants to only one of these symptom elicitation procedures.

SUMMARY:
College athletes will be recruited to complete a voluntary online survey that will take approximately 10 minutes. In this survey, they will answer a series of questions related to the concussion symptoms they have experienced in their recent sports season, their opinions related to concussions and concussion treatment, and demographics.

DETAILED DESCRIPTION:
College athletes will be recruited to complete a voluntary online survey that will take approximately 10 minutes. In this survey, they will answer a series of questions related to the concussion symptoms they have experienced in their recent sports season, their opinions related to concussions and concussion treatment, and demographics.

Of interest, participants will indicate what concussion symptoms they have recently experienced in one of four formats, to which they will be randomly assigned. Participants will either *check the symptoms they have experienced, *check the symptoms they have not experienced, *uncheck the symptoms they have experienced, or *uncheck the symptoms they have not experienced. It is believed that an alternative method of reporting symptoms that requires participants to indicate the symptoms they have not experienced will lead them to report having experienced a greater number of symptoms, based on past research regarding inclusion vs. exclusion modes of thought.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate athlete (identified by staff at each cooperating institution)

Exclusion Criteria:

* Under age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of symptoms | Through survey completion, an average of 12 minutes
  Participants are asked to indicate how many symptoms were experienced during their most recent sports season.

SECONDARY OUTCOMES:
Perceived risk of concussions | Through survey completion, an average of 12 minutes
  Using questionnaire, participants rate their perceived risk of having a concussion compared to the average American and the average college athlete over the next year.
Concern about concussions | Through survey completion, an average of 12 minutes
  Using questionnaire, participants rate their concern over having experienced a concussion in the past.
Concern about concussions for health | Through survey completion, an average of 12 minutes
  Using questionnaire, participants rate their concern about the risk concussions present to their health
Beliefs about responses to concussions | Through survey completion, an average of 12 minutes
  Using questionnaire, participants rate the extent to which they think others are concerned about concussions and should respond to concussions
Estimated number of concussions | Through survey completion, an average of 12 minutes
  Using questionnaire, participants estimate the number of concussions they experienced in the most recent sport season and in their life.
Knowledge about concussions | Through survey completion, an average of 12 minutes
  Using questionnaire, participants rate their own knowledge about concussions

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed by the research team and reported only in aggregate, so individual participant data will not be shared or made publicly available.